CLINICAL TRIAL: NCT00588549
Title: Utility of Whole-Body 18-Fluorodeoxyglucose Positron Emission Tomography (PET) In the Pre-Operative Assessment of Patients With Hepatic Colorectal Metastases
Brief Title: Utility of PET In the Pre-Operative Assessment of Patients With Hepatic Colorectal Metastases
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Yuman Fong, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 98-015
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to determine whether a test, called the PET scan, may be useful in determining if there are additional locations of cancer not otherwise detectable by other tests.

The PET scan is a nuclear medicine imaging study that measures how much radioactive sugar is used by your tumor. The study will compare pictures of the cancer from the PET scan to other x-ray exams, such as a CT scan, as well as to what your doctors find at the time of surgery. If the study results show that the PET scan gives us a good idea of what is happening to the tumor, then it may be useful in deciding which patients with colorectal metastases to the liver should be operated on and what operation should be performed.

Additionally, by comparing the results of PET scans with the other studies that will be performed as part of your care, we will try to determine which test best tells us which patient is most likely to benefit from surgery.

ELIGIBILITY:
Inclusion Criteria:

* initial diagnosis of colorectal carcinoma confirmed by the Pathology Department of Memorial Hospital or by diagnostic barium enema if the primary tumor is still in place.
* a candidate for liver resection for metastatic colorectal cancer as defined by members of the Department of Surgery of Memorial Hospital. Patients with metastatic colorectal cancer isolated to the colon, rectum, or liver are eligible. In addition, patients with limited, resectable pulmonary metastases are eligible.

Exclusion Criteria:

* Patients must not be pregnant; females of child bearing age must use an adequate form of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Memorial Sloan-Kettering Cancer Center patients with colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 1998-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess if whole body 18F-FDG-PET enhances our ability to detect metastatic colorectal cancer restricted to liver and lung over conventional imaging such as CT and to determine the accuracy of PET in imaging extrahepatic tumors. | conclusion of the study

SECONDARY OUTCOMES:
To determine whether PET plays a role in altering clinical management of patients undergoing evaluation for liver resection for hepatic colorectal metastases. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Yuman Fong, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm